CLINICAL TRIAL: NCT04480528
Title: The Effect of Various Strength Training Protocols in Female Runners With Patellofemoral Pain
Brief Title: Strength Training in Female Runners With Patellofemoral Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lauren Erickson (Other)
Collaborators: American College of Sports Medicine (Other)
Responsible Party: Sponsor-Investigator, Lauren Erickson, Graduate Research Assistant, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 54348
Record Dates: First submitted 2020-07-16; First posted 2020-07-21 (Actual); Last update posted 2022-03-04 (Actual); Status verified 2022-03

CONDITIONS: Patellofemoral Syndrome
Keywords: Blood Flow Restriction; Running; Patellofemoral Pain
MeSH Terms: conditions — Patellofemoral Pain Syndrome | interventions — Blood Flow Restriction Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BFRT Group (Experimental): This group will receive physical therapy plus active BFRT.
  Interventions: Other: Blood Flow Restriction Training (BFRT)
- Standard of Care Group (Sham Comparator): This group will receive physical therapy plus sham BFRT.
  Interventions: Other: Sham Blood Flow Restriction Training (Sham BFRT)

INTERVENTIONS:
Other: Blood Flow Restriction Training (BFRT) — A pressurized cuff is applied to the proximal thigh in order to partially occlude blood flow as the patient exercises.
  Arms: BFRT Group
Other: Sham Blood Flow Restriction Training (Sham BFRT) — A minimally pressurized cuff is applied to the proximal thigh in order to mimic the active blood flow restriction unit as the patient exercises.
  Arms: Standard of Care Group

SUMMARY:
Patellofemoral pain (PFP) is a common running-related injury that is often referred to as runner's knee. The condition typically presents with pain in the front of the knee that is located around or behind the knee cap. This injury occurs twice as frequently in females and is often associated with weakness of the muscles of the thigh and hip, as well as altered running form. Heavy-weight strength training is needed in order to improve muscle weakness; however, this puts a significant amount of load on the knee joint and it is difficult for individuals with PFP to train at this level without experiencing increased pain and joint discomfort. Blood flow restriction training (BFRT) is a promising alternative method to safely improve muscle weakness while reducing knee joint loading. With BFRT, a pressurized band is applied to the thigh in order to partially restrict blood flow as a patient exercises in order to decrease the amount of oxygen delivered to the muscle. Lack of oxygen to the muscle combined with strength training creates an environment within the muscle that results in the ability of low-weight strength training to provide the same results as heavy-weight strength training.

This study will evaluate how low-weight strength training with and without BFRT affects thigh and hip strength, and consequently pain, function, running ability, and running form in female runners with PFP. The hypothesis is that 10 weeks of low-weight strength training with BFRT will lead to greater thigh and hip strength, reduced pain, improved knee function, improved running ability, and improved running form compared to low-weight strength training without BFRT. The expected results will have a significant impact within the running community by providing a safe and effective treatment that increases strength and improves running form while reducing pain and joint loading. This will also have an impact on the larger field of sports medicine by providing an alternative method to improve strength, as well as improve function when heavy-weight strength training is not well tolerated or unsafe due to injury.

ELIGIBILITY:
Inclusion Criteria:

* Pain around (peripatellar) or behind (retropatellar) the patella, which is aggravated by running and at least one other activity that loads the patellofemoral joint during weight bearing on a flexed knee such as kneeling, squatting, stair ambulation, and jumping/hopping
* Insidious onset of symptoms unrelated to trauma
* Pain present for at least 2 months
* Pain rating of at least 3/10 on the visual analog scale during running
* Report running at least 10 miles per week currently or just prior to onset of injury
* Score a maximum of 85% on either the Knee Outcome Survey Activities of Daily Living Scale or Sports Activity Scale (KOS-ADL or KOS-SAS)

Exclusion Criteria:

* Knee pain resulting from acute trauma
* Concurrent ligamentous instability, meniscus pathology, patellar or iliotibial band tendinopathy
* History of patellar dislocations or instability, or previous reconstructive surgery to the knee
* Other lower extremity or lower back injury within the past 6 months

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2020-06-08 (Actual); Primary Completion 2021-11-13 (Actual); Study Completion 2021-11-13 (Actual)

PRIMARY OUTCOMES:
Change in Isometric Quadriceps Strength | 10 weeks
  The subject will be seated in a Biodex 4 dynamometer with their knee locked at 90 degrees of flexion. The subject will be asked to kick into the dynamometer pad as hard as they can and the peak force will be measured and normalized to body weight. Increased force indicates greater quadriceps strength.
Change in Isokinetic Quadriceps Strength | 10 weeks
  The subject will be seated in a Biodex 4 dynamometer and be asked to kick back-and-forth into the dynamometer pad as hard and as fast as they can. The peak force will be measured and normalized to body weight. Increased force indicates greater quadriceps strength.
Change in Isometric Hip Abduction Strength | 10 weeks
  The subject will be lying in the side-lying position with a stabilizing strap placed around the thigh. The subject will be asked to press out as hard as they can against a handheld dynamometer which records the force applied against it. The peak force will be measured and normalized to body weight. Increased force indicates greater hip abduction strength.
Change in Isometric Hip Extension Strength | 10 weeks
  The subject will be lying on their stomach with their knee flexed to 90 degrees and a stabilizing strap placed around the thigh. The subject will be asked to press up as hard as they can against a handheld dynamometer which records the force applied against it. The peak force will be measured and normalized to body weight. Increased force indicates greater hip extension strength.
Change in Isometric Hip External Rotation Strength | 10 weeks
  The subject will be seated with their knee flexed to 90 degrees and a stabilizing strap placed around the lower leg. The subject will be asked to press inward as hard as they can against a handheld dynamometer which records the force applied against it. The peak force will be measured and normalized to body weight. Increased force indicates greater hip external rotation strength.

SECONDARY OUTCOMES:
Change in Hip Adduction Angle | 10 weeks
  Change in peak hip adduction angle will be measured via a three-dimensional running gait analysis on an instrumented treadmill.
Change in Hip Internal Rotation Angle | 10 weeks
  Change in peak hip internal rotation angle will be measured via a three-dimensional running gait analysis on an instrumented treadmill.
Change in Peak Knee Extensor Moment | 10 weeks
  Change in peak knee extensor moment will be measured via a three-dimensional running gait analysis on an instrumented treadmill.
Change in Pain: Brief Pain Inventory (BPI) | 10 weeks
  Pain will be measured using the Brief Pain Inventory (BPI), which assesses pain (least, most, average, and present pain) on a scale from 0-10. Lower numbers indicate less pain while higher numbers indicate more pain.
Change in Patellofemoral Pain: Knee Injury and Osteoarthritis Outcome Score | 10 weeks
  Patellofemoral pain will be measured using the Knee Injury and Osteoarthritis Outcome Score - Patellofemoral Pain. It is an 11-item questionnaire and items are coded from 0 to 4, no problems to extreme problems. Scores are transformed to a 0-100 scale and represent the percentage of total possible score achieved. Lower numbers indicate greater knee patellofemoral pain while higher numbers indicate less patellofemoral pain.
Change in Knee Function | 10 weeks
  Knee function will be measured using the Knee Injury and Osteoarthritis Outcome Score (KOOS) which contains 5 subscales: Pain - 9 items, other Symptoms - 7 items, Function in daily living (ADL) - 17 items, Function in Sport and Recreation (Sport/Rec) - 5 items, and knee-related Quality of Life (QoL) - 4 items. Items are coded from 0 to 4, no problems to extreme problems. Scores are transformed to a 0-100 scale and represent the percentage of total possible score achieved. Lower numbers indicate greater knee problems while higher numbers indicate less knee problems.
Change in Running Ability | 10 weeks
  Running ability will be measured using the University of Wisconsin Running Injury and Recovery Index (UWRI). It is a 9-item questionnaire and items are coded from 0 to 4, lower scores indicating an inability to run and higher scores indicating no pain/issue with running. Scores are transformed to a 0-100 scale and represent the percentage of total possible score achieved. Lower numbers indicate limited running ability while higher numbers indicate full running ability.

CONTACTS AND LOCATIONS:
Overall Officials: Lauren Erickson, DPT, Principal Investigator — University of Kentucky
Locations (1):
- University of Kentucky, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No